CLINICAL TRIAL: NCT01277978
Title: Haemodynamic Assessment at Primary Caesarean Section After Administration of Carbetocin Versus Oxytocin: a Doubleblind Randomized Trail
Brief Title: Haemodynamic Effects of Oxytocin and Carbetocin
Status: Completed | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Manfred G. Mörtl, Dr. med., Medical University of Graz, Department of Obstetrics and Gynecology
Other Study IDs: CARBOXY-005498-78-Graz; 2007-005498-78 (EudraCT Number)
Record Dates: First submitted 2011-01-13; First posted 2011-01-17 (Estimated); Last update posted 2011-01-17 (Estimated); Status verified 2011-01

CONDITIONS: Pregnancy Related; Cesarean Section; Complications; Adverse Reaction to Oxytocic Agents
Keywords: Caesarean section; Cardiovascular effects; Postpartum hemorrhage; Carbetocin; Oxytocin
MeSH Terms: conditions — Postpartum Hemorrhage

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Carbetocin: Women undergoing elective caesarean sectio in regional anesthesia randomised to receive 100 ug Carbetocin (the clinical standard dose) following delivery of the baby.
- Oxytocin: Women undergoing elective caesarean sectio in regional anesthesia randomised to receive 5 IU oxytocin (the clinical standard dose) following delivery of the baby.

SUMMARY:
The purpose of this study is to evaluate the immediate effects of carbetocin and oxytocin on maternal hemodynamic parameters (heart rate and blood pressure) in a non-invasive setup (TaskeForce®-Monitor) during primary Caesarean section.

DETAILED DESCRIPTION:
As there is a trend toward childbearing in later life, pre-existing maternal cardiovascular problems may become more frequent during pregnancy and at delivery. In addition the increasing number of women with congenital or acquired cardiac diseases may not tolerate the induced haemodynamic changes as well as healthy patients. Therefore uterotonic drugs must be safe for the cardiovascular system.

Currently oxytocin is used as a common uterotonic agent in obstetrics. The use of this drug in uterotonic reasons can cause serious haemodynamic side effects which has been shown by several investigators.

Preliminary clinical observations of maternal heart rate and blood pressure suggest that that the use of carbetocin causes less hemodynamic changes than oxytocin.

Primary objective(s):

To evaluate the effect of carbetocin on maternal hemodynamic parameters (heart rate, blood pressure, systemic vascular resistance, cardiac output, stroke volume, heart rate variability, and blood pressure variability) in a non-invasive setup (TaskeForce®-Monitor) during primary Caesarean section.

To compare the haemodynamic changes of carbetocin versus oxytocin.

Secondary objective(s) To evaluate the need of additional drugs and methods to control uterine tone.

ELIGIBILITY:
Inclusion Criteria:

* Healthy pregnant women undergoing elective caesarean section with regional anesthesia

Exclusion Criteria:

---Women with

* placenta praevia
* placental abruption
* multiple gestation
* pregnancy related complications and disorders (i.e. preeclampsia, gestational diabetes)
* pre-existing diseases (e.g. insulin-dependent diabetes, cardiovascular or renal diseases, thyroid disease
* taking medication with known impact on the cardiovascular system
* undergoing caesarean section with general anesthesia
* secondary caesarean section

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women undergoing elective caesarean section after regional anesthesia at an University hospital providing intrapartum care.
Sampling Method: Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2008-01; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Immediate hemodynamic effects of carbetocin and oxytocin | 1 day
  Maternal heart rate, blood pressure, stroke volume, cardiac output, and systemic vascular resistance will be measured non-invasively.
  Measurements will be performed starting immediately following administration of the study medication.

SECONDARY OUTCOMES:
Adverse effects | 2 day
  Number of participants with adverse events as a measure of safety and tolerability
Uterotonic effect | 1 day
  Impact of both drugs on uterine tone
Estimation of blood loss | 2 day
  Measurement of pre- and postoperative hemoglobin levels (routine clinical blood sample).

CONTACTS AND LOCATIONS:
Overall Officials: Manfred G Mörtl, MD, Principal Investigator — Medical University Graz, Dept. of Obstetrics and Gynecology
Locations (1):
- Medical University Graz, Dept. of Obstetrics and Gynecology, Graz, Styria, Austria

REFERENCES:
- [Background] Pinder AJ, Dresner M, Calow C, Shorten GD, O'Riordan J, Johnson R. Haemodynamic changes caused by oxytocin during caesarean section under spinal anaesthesia. Int J Obstet Anesth. 2002 Jul;11(3):156-9. doi: 10.1054/ijoa.2002.0970. PMID 15321540
- [Background] Su LL, Chong YS, Samuel M. Oxytocin agonists for preventing postpartum haemorrhage. Cochrane Database Syst Rev. 2007 Jul 18;(3):CD005457. doi: 10.1002/14651858.CD005457.pub2. PMID 17636798
- [Background] Chong YS, Su LL, Arulkumaran S. Current strategies for the prevention of postpartum haemorrhage in the third stage of labour. Curr Opin Obstet Gynecol. 2004 Apr;16(2):143-50. doi: 10.1097/00001703-200404000-00008. PMID 15017343
- [Background] Westhoff G, Cotter AM, Tolosa JE. Prophylactic oxytocin for the third stage of labour to prevent postpartum haemorrhage. Cochrane Database Syst Rev. 2013 Oct 30;(10):CD001808. doi: 10.1002/14651858.CD001808.pub2. PMID 24173606
- [Background] Sweeney G, Holbrook AM, Levine M, Yip M, Alfredsson K, Cappi S, et al. Pharmacokinetics of carbetocin, a long-acting oxytocin analogue, in nonpregnant women. Curr Ther Res 1990;47:528-40
- [Background] Thomas JS, Koh SH, Cooper GM. Haemodynamic effects of oxytocin given as i.v. bolus or infusion on women undergoing Caesarean section. Br J Anaesth. 2007 Jan;98(1):116-9. doi: 10.1093/bja/ael302. Epub 2006 Dec 2. PMID 17142825
- [Background] Boucher M, Horbay GL, Griffin P, Deschamps Y, Desjardins C, Schulz M, Wassenaar W. Double-blind, randomized comparison of the effect of carbetocin and oxytocin on intraoperative blood loss and uterine tone of patients undergoing cesarean section. J Perinatol. 1998 May-Jun;18(3):202-7. PMID 9659650
- [Background] Dansereau J, Joshi AK, Helewa ME, Doran TA, Lange IR, Luther ER, Farine D, Schulz ML, Horbay GL, Griffin P, Wassenaar W. Double-blind comparison of carbetocin versus oxytocin in prevention of uterine atony after cesarean section. Am J Obstet Gynecol. 1999 Mar;180(3 Pt 1):670-6. doi: 10.1016/s0002-9378(99)70271-1. PMID 10076146
- [Background] Boucher M, Nimrod CA, Tawagi GF, Meeker TA, Rennicks White RE, Varin J. Comparison of carbetocin and oxytocin for the prevention of postpartum hemorrhage following vaginal delivery:a double-blind randomized trial. J Obstet Gynaecol Can. 2004 May;26(5):481-8. doi: 10.1016/s1701-2163(16)30659-4. PMID 15151735
- [Background] Atke A, Vilhardt H. Uterotonic activity and myometrial receptor affinity of 1-deamino-1-carba-2-tyrosine(O-methyl)-oxytocin. Acta Endocrinol (Copenh). 1987 May;115(1):155-60. doi: 10.1530/acta.0.1150155. PMID 3035851
- [Background] Hunter DJ, Schulz P, Wassenaar W. Effect of carbetocin, a long-acting oxytocin analog on the postpartum uterus. Clin Pharmacol Ther. 1992 Jul;52(1):60-7. doi: 10.1038/clpt.1992.103. PMID 1623693
- [Derived] Moertl MG, Friedrich S, Kraschl J, Wadsack C, Lang U, Schlembach D. Haemodynamic effects of carbetocin and oxytocin given as intravenous bolus on women undergoing caesarean delivery: a randomised trial. BJOG. 2011 Oct;118(11):1349-56. doi: 10.1111/j.1471-0528.2011.03022.x. Epub 2011 Jun 14. PMID 21668768